CLINICAL TRIAL: NCT05155072
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Pharmacokinetic/Pharmacodynamic Characteristics After Oral Administration of DW1903, DW1903-R1 and DW1903-R2 in Healthy Adult Volunteers
Brief Title: Clinical Trial to Evaluate the Safety and Pharmacokinetic/Pharmacodynamic Characteristics of DW1903
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW1903-101D
Record Dates: First submitted 2021-10-28; First posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-10

CONDITIONS: Gastritis
MeSH Terms: conditions — Gastritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence A (Experimental)
  Interventions: Drug: DW1903; Drug: DW1903-R1; Drug: DW1903-R2
- Sequence B (Experimental)
  Interventions: Drug: DW1903; Drug: DW1903-R1; Drug: DW1903-R2
- Sequence C (Experimental)
  Interventions: Drug: DW1903; Drug: DW1903-R1; Drug: DW1903-R2
- Sequence D (Experimental)
  Interventions: Drug: DW1903; Drug: DW1903-R1; Drug: DW1903-R2
- Sequence E (Experimental)
  Interventions: Drug: DW1903; Drug: DW1903-R1; Drug: DW1903-R2
- Sequence F (Experimental)
  Interventions: Drug: DW1903; Drug: DW1903-R1; Drug: DW1903-R2

INTERVENTIONS:
Drug: DW1903 — DW1903
Drug: DW1903-R1 — DW1903-R1
Drug: DW1903-R2 — DW1903-R2

SUMMARY:
A Randomized, Open-label, Oral in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers who are ≥19 years old
* BMI between 18 and 30 kg/m2
* Body weight ≥50kg

Exclusion Criteria:

•Clinically significant Medical History

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
pH monitoring | up to day 5
  Pharmacodynamic Endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, South Korea